CLINICAL TRIAL: NCT01776905
Title: In Vivo Real-time Detection of Circulating Melanoma Cells
Status: Recruiting | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 133965
Record Dates: First submitted 2013-01-14; First posted 2013-01-28 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Melanoma
Keywords: Melanoma; Cancer
MeSH Terms: conditions — Melanoma; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy control subjects: Characterize the baseline PA signals produced by the in vivo PAFC prototype device in healthy volunteers or Develop Standard Curves for the ex vivo CTC assays.
- Advanced-Stage Melanoma: To validate the in vivo PAFC method of melanoma CTC detection, we will use the PAFC-based prototype device to noninvasively determine CTC concentrations in the blood of subjects who have advanced-stage (Stage III or Stage IV)melanoma, and we will also use current ex vivo methods to determine the CTC concentration in samples of blood drawn from the same subjects.
- Early-Stage Melanoma: To determine whether in vivo PAFC can detect melanoma CTCs at concentrations below the detection limits of the ex vivo methods, we will use the PAFC-based prototype device to noninvasively detect CTCs in the blood of subjects who have early-stage (Stages I or II) melanoma, and we will also use current ex vivo methods to detect CTCs in samples of blood drawn from the same subjects.

SUMMARY:
The objective of this clinical trial is to determine whether a Photoacoustic flow cytometry (PAFC)-based prototype device can detect circulating tumor cells (CTCs) in the blood of melanoma patients in vivo, in real time, and do so at detection limits at least one order of magnitude below the detection limits of currently existing ex vivo methods.

DETAILED DESCRIPTION:
Study Population: Approximately 80 subjects will be consented in order to achieve an enrollment goal of 75 subjects at this institution in three cohorts as follows:

1. Cohort #1 will consist of fifteen healthy control subjects, ten of whom will be Caucasian and five of whom will be African-American. Subjects in cohort #1 will be used to address the calibration goal of Specific Aim #1.
2. Cohort #2 will consist of 30 subjects who have advanced-stage melanoma will be recruited from the Medical Oncology clinic at UAMS, where advanced stages are defined as Stages III or IV. Subjects in cohort #2 will be used to address the validation goal of Specific Aim #2. Approximately half of the 30 advanced-stage subjects will be Stage III and the other half will be Stage IV.
3. Cohort #3 will consist of 30 subjects with early-stage melanoma will be recruited from the Surgical Oncology clinic at UAMS, where early stages are defined as Stages I or II.

Subjects in cohort #3 will be used to address the detection goal of Specific Aim #3. Approximately 10 of the 30 early-stage subjects will be Stage I and approximately 20 will be Stage II.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years
* Histological documented diagnosis of melanoma
* Signed informed consent form approved by the University of Arkansas for Medical Sciences (UAMS) Institutional Review Board (IRB)
* Must be able to sit still for 90 minutes

Exclusion Criteria:

* Active infection
* Current and significant medical or surgical condition as determined by the Investigator
* Diagnosis or evidence of organic brain syndrome
* Pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Expect to consent approximately 80 subjects in order to achieve an enrollment goal of 75 subjects at this institution in three cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants that possess circulating tumor cells. | 14-21 days

CONTACTS AND LOCATIONS:
Overall Officials: Jumin Sunde, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States